CLINICAL TRIAL: NCT01146548
Title: Assessment of Fluoxetine's Effect in Patients With Multiple System Atrophy : a Double Blind Placebo-controlled Randomized Trial
Brief Title: Fluoxetine in Multiple System Atrophy Patients
Acronym: MSA-Fluox
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Clinical Research Center, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 0720101
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2012-02

CONDITIONS: Multiple System Atrophy
Keywords: Fluoxetine effect; Multiple System Atrophy; MSA
MeSH Terms: conditions — Multiple System Atrophy | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- the fluoxetine group (Experimental): Multiple System Atrophy's patients with fluoxétine
  Interventions: Drug: FLUOXETINE
- the placebo group (Placebo Comparator): Multiple System Atrophy's patients with placebo
  Interventions: Drug: FLUOXETINE

INTERVENTIONS:
Drug: FLUOXETINE — 20mg/d, oral administration for 6 weeks, then 40mg/d for 4 months.
  Other Names: PROZAC®

SUMMARY:
This is a French national trial, conducted using a double-blind, placebo-controlled, randomised design involving 15 centers and 88 patients of both sexes.

The primary objective of the trial is to evaluate the effect of a selective inhibitor of serotonin reuptake, the Fluoxétine, at a higher dose (40 mg/day) than usually recommended for depressed patients, after three months in patients suffering from an atypical Parkinson's disease called Multiple System Atrophy, compared to the placebo effect.

Secondary objectives of the trial are the evaluation of the effects of Fluoxétine after six weeks at the dose of 20 mg/day, after six months at the dose of 40mg/day, and assess the effects on mortality, quality of life, autonomic disorders, particularly orthostatic hypotension, mood and others symptoms such as sleep, apathy, pain and fatigue.

DETAILED DESCRIPTION:
Fluoxetine is first introduced in dose of 20 mg/day and after six weeks the dose is increased to 40 mg/day. If patients have side effects at the dose of 40 mg/day, the dose may be reduced at 20 mg/day. Assessment visits will be conducted at 6 weeks, 3 months, and 6 months of treatment. After 6 months, trial's treatment with fluoxetine is discontinued gradually. A new assessment will be conducted one month after the end of treatment. The expected results are the demonstration of improved scores of the scale UMSARS after 3 and 6 months in the fluoxetine group compared to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Female or Male Patient with Multiple System Atrophy's disease diagnosed according to international consensus criteria (Gilman's criteria)
* Patient between 30 and 80 years of age
* Patient not presenting a cognitive problem that could impair the comprehension of the patient and his participation in the protocol
* Patient receiving an anti-parkinsonian treatment (if applicable) at a stable dose for at least 2 months before entering the study, and with the expectation that the treatment will remain unchanged throughout the course of the patients participation in the trial
* Patient receiving a symptomatic treatment of autonomic disorders (if applicable) at a stable dose for at least 2 months before entering the study, and with the expectation that the treatment will remain unchanged throughout the course of the patient participation in the trial
* Signed informed consent obtained
* Patient eligible for social security (specific requirement under French law)

Exclusion Criteria:

* Patient presenting major swallowing problems as he will not take capsule
* Patient already receiving a selective inhibitor of serotonin reuptake or other antidepressant, or patient having received one in the 3 months preceding the start of the study
* Patient with major depressive syndrome for which the investigator considers that the indication of an antidepressant seems essential
* Bedridden patient or confined to a wheelchair during the whole day
* Patient with severe hyponatremia
* Patient with another Parkinsonian's syndrome that the Multiple System Atrophy (type of atypical Parkinson's disease, progressive supra nuclear paralysis, cortico-basal degeneration)
* Patient with dementia
* Patient with a Mini-Mental State Exam score < 24
* Patient unable to understand the protocol or another endpoint or to consider the clinical trial's process
* Patient with a chronic disease affecting the development or assessment of the patient during the trial
* Patient receiving concomitant medications which could affect the evaluation of outcome measures (e.g. neuroleptics for the assessment of parkinsonian symptoms, vasodilators for the assessment of orthostatic hypotension, sedative drugs prescribed during the day for the assessment of the daytime sleepiness, of apathy or of fatigue)
* Patient with absolute or relative contraindications of Fluoxetine (hypersensitivity to Fluoxetine, patient with a history of epilepsy, of manic state, of severe hepatic or renal impairment, of skin bleeding, of severe heart, of uncontrolled diabete, patient treated by selective or non selective IMAO)
* Person who are: wards of the state or prisoners (requirement under french law)
* Patient pregnant or at risk of same, nursing mother

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2008-05; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
primary efficacy endpoint | 3 months
  The primary efficacy endpoint is the comparison of scores in Parts I and II of the UMSARS scale between the visit V0 and V2 (i.e. after 3 months of treatment at the dose of 40mg/day).

SECONDARY OUTCOMES:
secondary efficacy endpoints | 6 weeks, 3 months or 6 months
  * comparison of scores in Parts I and II of the UMSARS scale between the visit V0 and V3, i.e. after 6 months of treatment at the dose of 40mg/d
  * comparison of scores in Parts I and II of the UMSARS scale between the visit V0 and V1, i.e. after 6 weeks of treatment at the dose of 20mg/d
  * rate of mortality
  * score of SCOPA AUT scale - assessment of symptomes related to the dysautonomic affect
  * score of Part III of UMSARS scale - assessment of orthostatic hypotension
  * score of Beck scale - assessment of depression
  * score of Schrag scale - assessment of health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Rascol, MD, Principal Investigator — Hospital University Toulouse
Locations (14):
- France (14):
  - Hospital, Nantes, France
  - hospital center of Aix enProvence, Aix-en-Provence
  - Hospital Gabriel Montpied, Clermont-Ferrand
  - University Hospital Henri Mondor, Créteil
  - Hopital, Dijon
  - Hospital R Salengro, Lille
  - university hospital Dupuytren, Limoges
  - university hospital Timone, Marseille
  - University Hospital, Montpellier
  - hospital Pitié Salpêtrière, Paris
  - University Hospital La Miletrie, Poitiers
  - Hospital Pontchaillou, Rennes
  - civil hospital of Strasbourg, Strasbourg
  - University Hospital, Toulouse